CLINICAL TRIAL: NCT01019083
Title: Studies of Acute and Memory Immune Responses to Orally Administered Vaccines in Developing Country Children and Factors That May Augment Such Responses
Brief Title: Studies of Immune Responses to Orally Administered Vaccines in Developing Country
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: International Centre for Diarrhoeal Disease Research, Bangladesh (Other)
Collaborators: Göteborg University (Other)
Responsible Party: Dr. Firdausi Qadri, International Centre for Diarrhoeal Disease Research, Bangladesh
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Basic Science
Other Study IDs: 2007-066
Record Dates: First submitted 2009-11-22; First posted 2009-11-25 (Estimated); Last update posted 2011-07-12 (Estimated); Status verified 2009-11

CONDITIONS: Cholera; Typhoid
Keywords: Cholera; Typhoid; Oral Vaccine; Immune response; Vaccine Evaluation; Nutrition; Child Health
MeSH Terms: conditions — Cholera; Typhoid Fever | interventions — Zinc Sulfate; Albendazole; secnidazole; Arsenic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- zinc supplementation-Placebo (Placebo Comparator): Determine if the immunogenicity of oral typhoid can be enhanced in children by introducing zinc supplementation: Our recent studies on the interactions of oral cholera vaccine with breast milk and zinc provide some basis for improving immunogenicity, but additional work is needed to improve many of the oral vaccines. In this study we also plan to evaluate if the immune response to Cholera and Vivotif can be enhanced by supplementation with zinc using methods described earlier. We would like to study children, 2-5 years of age for this purpose.
  Interventions: Drug: Placebo
- Anti Parasite Drug- Placebo (Placebo Comparator): There is a high burden of enteric parasites in the gut of people living in densely populated areas of less developed countries. The effect of concurrent parasitic infestations on immune responses has not been studied widely, although it is an area of utmost importance for natural protection as well as vaccine immuno-prophylaxis. In this study we plan to determine the impact of pretreatment with antiparasitic agents (albendazole and secnidazole) on the immunogenicity of the oral cholera and typhoid vaccines in children, 2-5 years of age
  Interventions: Drug: Placebo
- Effect of Arsenic in Dukoral- Control (Experimental): In this study, we aim to evaluate if immunogenicity of the oral cholera vaccine is modified in children living in a high arsenic contaminated area in Bangladesh. The plan is to study children 2-5 year old living in Shahrasti thana near Matlab where the tubewell water is highly contaminated with arsenic and this study will not be randomized double-blind, and compare their responses with responses of age matched children living in arsenic free area, such as in Mirpur area of Dhaka city. We only plan to study the effect of Dukoral vaccinees since this vaccine has been widely studied in Bangladesh. If an impact of arsenic is seen on immune response to this vaccine, future studies could be done with other vaccines including Vivotif.
  Interventions: Other: Control
- zinc supplementation (Experimental): Determine if the immunogenicity of oral typhoid can be enhanced in children by introducing zinc supplementation: Our recent studies on the interactions of oral cholera vaccine with breast milk and zinc provide some basis for improving immunogenicity, but additional work is needed to improve many of the oral vaccines. In this study we also plan to evaluate if the immune response to Cholera and Vivotif can be enhanced by supplementation with zinc using methods described earlier. We would like to study children, 2-5 years of age for this purpose.
  Interventions: Drug: Zinc Sulphate
- administration of antiparasitic drugs (Experimental): There is a high burden of enteric parasites in the gut of people living in densely populated areas of less developed countries. The effect of concurrent parasitic infestations on immune responses has not been studied widely, although it is an area of utmost importance for natural protection as well as vaccine immuno-prophylaxis. In this study we plan to determine the impact of pretreatment with antiparasitic agents (albendazole and secnidazole) on the immunogenicity of the oral cholera and typhoid vaccines in children, 2-5 years of age
  Interventions: Drug: Albendazole and Secnidazole
- Effect of arsenic on Dukoral response (Experimental): In this study, we aim to evaluate if immunogenicity of the oral cholera vaccine is modified in children living in a high arsenic contaminated area in Bangladesh. The plan is to study children 2-5 year old living in Shahrasti thana near Matlab where the tubewell water is highly contaminated with arsenic and this study will not be randomized double-blind, and compare their responses with responses of age matched children living in arsenic free area, such as in Mirpur area of Dhaka city. We only plan to study the effect of Dukoral vaccinees since this vaccine has been widely studied in Bangladesh. If an impact of arsenic is seen on immune response to this vaccine, future studies could be done with other vaccines including Vivotif.
  Interventions: Other: Arsenic

INTERVENTIONS:
Drug: Placebo — Placebo will be given according to randomization list
  Other Names: Zinc Sulphate
  Arms: zinc supplementation-Placebo
Drug: Placebo — Placebo will be given according to randomization list
  Other Names: Albendazole and Senidazole
  Arms: Anti Parasite Drug- Placebo
Other: Control — Control will be selected from the Arsenic non contaminated Area
  Other Names: Arsenic Contaminated Area
  Arms: Effect of Arsenic in Dukoral- Control
Drug: Zinc Sulphate — Zinc Sulphate will be given according to randomization list
  Other Names: Placebo
  Arms: zinc supplementation
Drug: Albendazole and Secnidazole — Albendazole and Secnidazole will be given according to randomization list
  Other Names: Placebo
  Arms: administration of antiparasitic drugs
Other: Arsenic — Participant will be selected from the Arsenic Contaminated Area
  Other Names: Non contaminated Arsenic area
  Arms: Effect of arsenic on Dukoral response

SUMMARY:
The efficacy and immunogenicity of enteric vaccines have generally been found to be lower in children in the developed than in the developing countries. This has been observed with vaccines against cholera rotavirus, ETEC and typhoid vaccines. There are a number of factors that may contribute to such differences in vaccine "take rates" in children, e.g. breast feeding and nutritional status of the children might influence their immunogenicity and efficacy. Thus, breast feeding of newborn and young infants may adversely influence the immune response to vaccination, which might have more pronounced effect in developing than in developed countries. Breastfeeding has also been shown to interfere with the serum immune responses to rotavirus vaccine although this effect could be overcome by administering three rather than one dose of the oral rotavirus vaccine. Our recent study of Dukoral in Bangladeshi children aged 18 months or younger has shown that the response rates and the magnitude of responses improved when breast milk was temporarily withheld . Thus, administration of vaccines may have to be adjusted when given to breast fed children. Another factor that may affect the immunogenicity is the effect of zinc. Previous studies have shown that zinc enhances the immune response to cholera vaccine in participants > 2 years of age , a recent study also observed a similar effect in infants.

In this research project, we plan to study a number of different factors that might influence the immunogenicity of the two licensed oral model vaccines, specifically the inactivated killed oral cholera vaccine, Dukoral, and the live oral typhoid vaccine, Ty21a. We will also identify strategies that might improve the immunogenicity of the vaccines. The main objective of our study is to identify immunization regimens that may improve the immunogenicity of the vaccines in young children, which could be subsequently in field trials in Bangladesh and other developing countries. Specifically, we will determine if: (i) interventions identified to enhance immune responses to Dukoral, including zinc supplementation, could also enhance the immune responses to Ty21a; (ii) these two vaccines are able to induce both acute and memory B and T cell responses, (iii) treatment with antiparasitic drugs prior to immunization could modulate the immune responses to cholera and typhoid vaccines; and (iv) examine if arsenic exerts a suppressive effect on the immunogenicity of these vaccines.

DETAILED DESCRIPTION:
Research Design and Methods

Vaccine field sites and overall study design:

Mirpur. The vaccine studies will be carried out at the field site in Mirpur, in urban Dhaka, where oral cholera, ETEC and rotavirus studies as well as amoebiasis studies are being conducted over the last 15 years . For the Dukoral vaccine, two doses will be given to the study participants, 14 days apart. In case of Vivotif, 3 doses will be administered on alternate days i.e. days 1, 3 and 5 or in two doses 28 days apart.

Blood and stool samples will be collected prior to vaccination, and 7 days after intake of each dose of the cholera vaccine and 7 days after the intake of last dose of typhoid vaccine, and the volumes to be sampled for immunological assays have been described in Appendix 2. The participants will not be allowed to eat or drink from one hour before and one hour after intake of the vaccine. To assess the effect of zinc on immune response to typhoid vaccine in young children, supplementation will be initiated 2 weeks before the first dose and will continue up to 21 days after the last (third) dose of typhoid vaccine (that is for a total of 40 days).

Serum zinc concentrations will be determined at baseline only. Venous blood will be collected in trace element free vacutainers, which will be placed in ice until arrival at the ICDDR,B laboratory the same day.

Vaccine studies in an arsenic contaminated area in Shahrasti:

Shahrasti thana with a population of around 200,000 is located about 40 kilometers from Matlab, and is well connected with Comilla, Chandpur and Dhaka by road. According to BAMWSP (Bangladesh Arsenic Mitigation Water Supply Project), subsoil water in Shahrasti Thana is heavily contaminated with arsenic; about 99% of the tube wells are reported to have been contaminated (50 microgram/L). BAMWSP and DGHS have already identified 3000 patients with skin lesions consistent with arsenic toxicity, and represent the area with the second highest number of arsenic-induced skin lesions in Bangladesh. In collaboration with ICDDR,B, the University Chicago and Columbia University are jointly conducting a large longitudinal surveillance and clinical trial on patients with arsenic induced skin lesion. The aim of this large study is to reduce skin cancer by evaluating clinical as well biochemical markers. We plan to study responses of children in these sites to Dukoral using the infrastructure and facilities from the ongoing studies . The immunogenicity studies will be carried out as described earlier. We plan to immunize 102 children aged 2-5 years with two doses of Dukoral at an interval of 14 days. Equal numbers of children will be studied in an area known to have low levels of arsenic, in Mirpur field site in Dhaka city . This will be the first study to compare immune responses to a mucosal vaccine in an arsenic prone and arsenic low area.

Informed consent and selection of study subjects for vaccine studies:

Voluntary written informed consent will be obtained from the parent/guardians for participation of children including their vaccination and sampling of blood and stool for various assays (Appendices). Healthy children (1 - 5 years) and adults (18-45 years) both males and females living in the Mirpur field site, who are not currently enrolled in any other research study, whether conducted by ICDDR,B or other organization, will be screened and enrolled subject to meeting the eligibility criteria. Similar procedures will be followed for part of the Dukoral study that will be conducted in Shahrasti.

We have previously experienced that at least 60% of the families do agree to participation of their children in research studies. The prospective participants of this study will be carefully examined and assessed by a physician before enrollment. A detailed history of their previous immunizations will be obtained, and their nutritional status and recent illness (as outlined below) that could compromise the immune system and family background etc. will be considered before study enrollment. The participants should be free from any chronic disease or any recent illness that may compromise the immune system including arsenic related skin lesions in children in Shahrasti where only Dukoral vaccine would be evaluated.

Children will also be excluded if they have: (i) history of chronic gastrointestinal disorder; (ii) diarrheal illness in the past 2 weeks (diarrhea defined as passage of 3 or more abnormally loose or watery stool in a 24 hour period; (iii) any febrile illness in the preceding week; (iv) other chronic illness; (v) history of receiving antibiotic treatment within the last 7 day; and (vi) severe protein energy malnutrition (PEM). The nutritional status of the children will be assessed using anthropometric measurements (weight-for-age, and weight-for-length/height); children below -2SD for weight for height/length of the NCHS median will not be enrolled. Similarly, children who have received zinc in the past two months will also not be recruited.

Baseline laboratory assessments:

Stool: Microscopic examination, and culture for isolation and identification of enteric pathogens including ETEC. V. cholerae and S.Typhi will be carried out for four days prior to vaccination. Children who have any of these pathogens isolated from their stool specimen will not be vaccinated since they will confound evaluation of the response to the vaccine. When immunization for the second dose of the vaccine will be carried out (14 days after the first dose) children who have fever or diarrhea will be excluded from the study.

For arsenic related studies, urine will be collected and stored for assessment of levels of arsenic. This will be carried out in the Biochemistry and Nutrition Unit of ICDDR,B using standard procedures.

Vaccine, administration and allocation:

Dukoral. The cholera vaccine, Dukoral is produced by the Swedish Bacteriological Laboratories (SBL Vaccin AB Stockholm, Sweden). This inactivated, oral cholera vaccine consists of killed bacteria prepared from individual strains of O1 ElTor and classical V. cholerae that include both LPS and protein antigens, and also contains recombinant B subunit of cholera toxin (rCTB). One dose of vaccine contains 1.25 x 1011 killed whole cells plus 1 mg of rCTB. Immediately before use, individual doses of the liquid form of the vaccine will be mixed with the reconstituted bicarbonate buffer. For children, the vaccine will be suspended in 20 ml (total 4 teaspoon) of bicarbonate-citric acid buffer [the buffer is prepared by adding 100 ml water to a sachet of bicarbonate buffer (2 g bicarbonate; 750 mg of citric acid; Recip AB, Stockholm). For adults, Dukoral will be reconstituted in 100 ml of the buffer.

Vivotif: Live, attenuated oral typhoid vaccine, Vivotif, contains 2-6x109 CFU (colony-forming units) of S. Typhi Ty21a strain (1,2). The Berna Biotech Ltd, Berne, Switzerland, manufactures this vaccine. The enteric-coated, typhoid vaccines are packaged as sets of 3-capsules. The vaccine capsule is swallowed with drinking water and administered on alternate days i.e. days 1, 3 and 5. For immunization of children under 5 years of age, we plan to administer the vaccine in bicarbonate buffer as is the procedure in for children in travelers clinics (Sweden and USA). For this purpose the capsule is opened up and the contents suspended in 20 ml of bicarbonate buffer and then taken orally.

Overall sample size calculations:

The sample size has been estimated for different interventions, using a one-sided hypothesis with 95% confidence, a minimum detectable mean difference (DMD) of 50% improvement over the baseline, adjusted for around 15% dropouts.

In earlier Dukoral cholera vaccine studies in Bangladesh, 56% of the recipient children aged 6 months to 2 years responded with vibriocidal antibodies ; For the Vivotif vaccine data from vaccines aged >6 years documented 67% seroconversion. The sample sizes for different components of the study have been calculated based on the assumption that 50% of children will respond to Vivotif. Based on the results obtained with zinc supplementation on the immune response to Dukoral, that observed increase in the rates with supplementation from 56% to 79% , and assuming a 30% increase in responses to Vivotif (with around 15 attrition rates) the sample size will be 75 in each group (with and without zinc).

Prevalence of major enteric parasites in children 2-5 years of age in urban Dhaka is around 78%. To see the effects of anti-parasitic drug therapy prior to cholera and typhoid vaccination, we will enroll 102 children in each group in Dukoral (n=102x2=204) and and another 102 children in each group for Vivotif vaccine (102 x 2 = 204). For each vaccine, one group will be treated while another will not be. Thus we plan to study a total of 408 children to determine effect of anti-parasitic drugs on the immune responses to oral cholera and typhoid vaccines.

To determine the effect of arsenic on the immune response to Dukoral, we assume that the immunogenicity of the vaccine among children in the arsenic non-contaminated area will be 55% and in the contaminated area it will be reduced to 35%. To detect this difference with 95% confidence and 90% power, we estimated a sample size of 138 in each of the two study areas. With around 10% loss to follow up the required sample size will be 154. Thus, a total of 308 (154 x 2 = 308) children, aged 2-5 years, will be enrolled.

To determine the acute and memory B and T cell responses to oral cholera vaccine, studies will be conducted in adults (18-45 years) and children of different age groups (1 -5 years). For this part of the study, 25 adults, 25 toddlers (2-5 years old), and 25 under-two children will be vaccinated. For responses to Vivotif, we will only study adults (n=25) and toddlers (n-25).

The participants will be studied and followed up for the T and B cell responses prior to immunization, and during early post-immunization period (post- 7 days), and on 30 days, and 6, 12 and 24 months following the last dose.

Administration of associated interventions

Effect of zinc on the immune responses to Vivotif We would like to study the effect of zinc on the immunogenicity of oral typhoid vaccine and cholera vaccine by supplementing children with daily zinc sulfate (20 mg/day) for two weeks prior to immunization and until the last follow-up for sample collection (n=150).

Effect of anti-parasitic drugs on the immune responses to Vivotif and Dukoral A total 408 children will be enrolled to see the effects of anti parasitic therapy prior to cholera and typhoid vaccination, equal cholera and typhoid. For this purpose children will be given albendazole (400 mg) and secnidazole (500 mg) one week prior to immunization .

Study the effect of arsenic on the immune response to Dukoral This study will be conducted on children (2-5 years) in arsenic contaminated area (Shahrasti) and arsenic free area (Mirpur). For this purpose, a total of 308 children (154 from each site) will be enrolled and vaccinated with Dukoral. This study will for the first time compare immune responses to a mucosal vaccine in an arsenic prone and arsenic low area. Urine will be collected from all participants, prior to immunization for determining arsenic levels.

Determine the acute and memory B and T cell responses to oral cholera and typhoid vaccine in children and adults:

A total of 150 subjects will be vaccinated and followed up for T and B cell responses over a period during the early post-immunization period (7 days post-), 30 days, 6, 12 and 24 months later.

ELIGIBILITY:
Inclusion Criteria:

1. voluntary written informed consent will be obtained from the parent/guardians for participation of children including their vaccination and sampling of blood and stool for various assays.
2. healthy children (1 - 5 years)and adults (18-45 years) both males and females living in the Mirpur field site, who are not currently enrolled in any other research study, whether conducted by ICDDR,B or other organization, will be screened and enrolled subject to meeting the eligibility criteria. For Dukoral study that will be conducted in Shahrasti we will recruit only 2-5 years old children.

Exclusion Criteria:

1. history of chronic gastrointestinal disorder.
2. diarrheal illness in the past 2 weeks (diarrhea defined as passage of 3 or more abnormally loose or watery stool in a 24 hour period.
3. any febrile illness in the preceding week.
4. other chronic illness.
5. history of receiving antibiotic treatment within the last 7 day.
6. severe protein energy malnutrition (PEM). The nutritional status of the children will be assessed using anthropometric measurements (weight-for-age, and weight-for-length/height); children below -2SD for weight for height/length of the NCHS median will not be enrolled. Similarly, children who have received zinc in the past two months will also not be recruited.

Ages: 1 Year to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 1016 (Estimated)
Dates: Start 2008-02; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Determine if the immunogenicity of typhoid (Vivotif) and cholera vaccine (Dukoral) in young children is influenced by the factors i. zinc supplementation ii. antiparasitic drugs and iii. relationship between serum arsenic and immune response to Dukoral | 3 years

SECONDARY OUTCOMES:
Determine the acute and memory B and T cell responses to oral cholera and typhoid vaccine in children and adults | 3 Years

CONTACTS AND LOCATIONS:
Overall Officials: Firdausi Qadri, PhD, Principal Investigator — International Centre for Diarrhoeal Disease Research, Bangladesh
Locations (1):
- Firdausi Qadri, Dhaka, Bangladesh

REFERENCES:
- [Background] Qadri F, Ahmed T, Wahed MA, Ahmed F, Bhuiyan NA, Rahman AS, Clemens JD, Black RE, Albert MJ. Suppressive effect of zinc on antibody response to cholera toxin in children given the killed, B subunit-whole cell, oral cholera vaccine. Vaccine. 2004 Jan 2;22(3-4):416-21. doi: 10.1016/j.vaccine.2003.07.005. PMID 14670323
- [Background] Ahmed T, Svennerholm AM, Al Tarique A, Sultana GN, Qadri F. Enhanced immunogenicity of an oral inactivated cholera vaccine in infants in Bangladesh obtained by zinc supplementation and by temporary withholding breast-feeding. Vaccine. 2009 Feb 25;27(9):1433-9. doi: 10.1016/j.vaccine.2008.12.036. Epub 2009 Jan 13. PMID 19146904